CLINICAL TRIAL: NCT03039465
Title: A Novel Modified Tracheo-Esophageal Voice Prosthesis for Total Laryngectomy Patients
Acronym: TEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthCare Global Enterprise Ltd. (Industry)
Responsible Party: Principal Investigator, Vishal U S Rao, Head, Dept of Head & Neck Surgery, HealthCare Global Enterprise Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCG/SX/003/2016
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Laryngeal Cancer; Hypopharynx Cancer
Keywords: Indwelling Trachea-oesophageal Prosthesis; Voice Rehabilitation; Total Laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: A single group of patients undergoing the insertion of the prosthesis would be evaluated for voice quality and fluid leak as a measure of success of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Trans-Esophageal Prosthesis (Experimental): Patients satisfying the selection criteria would be subjected to the insertion of the TEP and evaluated at subsequent time points for the success of the procedure.
  Interventions: Device: Modified Trans-Esophageal Prosthesis

INTERVENTIONS:
Device: Modified Trans-Esophageal Prosthesis — This device is a biomedical grade silicon voice prosthesis with an inner esophageal flange, a stem and an outer tracheal flange. Insertion would be done through a modified 'romovac' inserter set / curved metal inserter (provided with the TEP) and an oesophagoscope in case of secondary insertion would be used. in patients with existing TEP puncture / who require a TEP change, on out-patient basis, the insertion would be done with a novel two-part inserter device (front loading)

SUMMARY:
This study is being conducted at Healthcare Global Enterprises Ltd to evaluate the role of a novel Tracheo-Esophageal voice Prosthesis for total laryngectomy +/- partial pharyngectomy patients. 30 patients will be enrolled as an inpatient or outpatient.

Patients who are planned to undergo total laryngectomy +/- pharyngectomy surgery and trachea-esophageal puncture procedure.(for primary TEP insertion) or patients who have undergone total laryngectomy > 6weeks prior and are suitable candidates for secondary TEP insertion would be recruited to the study. Insertion of the TEP will be done in primary setting or secondary setting. Patients, who are undergoing primary TEP insertion, will be evaluated for speech/ voice at an interval of 6 weeks, 12 weeks and 6 months after the procedure. Patients who are undergoing secondary TEP insertion to be evaluated on the same day of the procedure along with evaluation at an interval of 6 weeks, 12 weeks and 6 months. All the patients will be evaluated clinically for a fluid leak (through and around the TEP) on the same days of voice analysis by giving test feeds under supervision.

DETAILED DESCRIPTION:
This study is being conducted at Healthcare Global Enterprises Ltd to evaluate the role of a novel trachea-oesophageal prosthesis for total laryngectomy +/- partial pharyngectomy patients. 30 patients will be enrolled as an inpatient or outpatient.

Patients who are planned to undergo total laryngectomy +/- pharyngectomy surgery and trachea-esophageal puncture procedure.(for primary TEP insertion) or patients who have undergone total laryngectomy > 6weeks prior and are suitable candidates for secondary TEP insertion would be recruited to the study. Insertion of the TEP will be done in primary setting or secondary setting. Patients, who are undergoing primary TEP insertion, will be evaluated for speech/ voice at an interval of 6 weeks, 12 weeks and 6 months after the procedure. Patients who are undergoing secondary TEP insertion to be evaluated on the same day of the procedure along with evaluation at an interval of 6 weeks, 12 weeks and 6 months. All the patients will be evaluated clinically for fluid leak (through and around the TEP) on the same days of voice analysis by giving test feeds under supervision.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are surgically and medically fit for undergoing a total laryngectomy +/- partial pharyngectomy.
* Patients who have already undergone total laryngectomy +/- partial pharyngectomy and are willing for a secondary voice rehabilitation procedure.
* Patient signing the informed consent for procedure after understanding the details

Exclusion Criteria:

* Partial laryngectomy
* Near total laryngectomy
* Patient unfit for the procedure
* Patients not consenting for the procedure
* Patients utilizing alternative ways of post laryngectomy voice rehabilitation (for secondary insertion)
* Patients with stricture in pharynx (for secondary insertion)
* Partial pharyngectomy reconstruction, not permitting insertion of TEP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Voice Quality | Assessments would be done 6 weeks, 12 weeks and 6 months post surgery
  Voice quality would be assessed by a speech therapist using a standardized questionnaire to assess the functionality of the modified TEP
Change in Presence / Absence of Fluid Leak | Immediately, 6 weeks, 12 weeks and 6 months after the Modified TEP insertion procedure
  Clinical assessment of modified TEP leak after a test fluid feed

CONTACTS AND LOCATIONS:
Overall Officials: Vishal US Rao, MS, Principal Investigator — Dept of Head & Neck Surgery, HealthCare Global Enterprises Ltd.
Locations (1):
- HealthCare Global Enterprises Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Overall results of the study would be made public but individual patient data would be not be made available